CLINICAL TRIAL: NCT01023477
Title: Preventing Invasive Breast Neoplasia With Chloroquine (PINC) Trial
Brief Title: Study of the Efficacy of Chloroquine in the Treatment of Ductal Carcinoma in Situ (The PINC Trial)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: George Mason University (Other); University of Pittsburgh Medical Center (Other); United States Department of Defense (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFHCC 09-002
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-05

CONDITIONS: Carcinoma, Intraductal, Noninfiltrating; DCIS; Ductal Carcinoma In Situ
Keywords: Carcinoma, Intraductal, Noninfiltrating; Ductal Carcinoma In Situ; DCIS; Carcinoma, Intraductal; Breast Cancer; Breast Tumors; chloroquine; autophagy; Autophagic Cell Death; Autophagocytosis; Programmed Cell Death, Type II; Autophagy, Cellular; Autophagic Programmed Cell Death
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms | interventions — Chloroquine; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chloroquine Standard Dose (500mg/week) (Experimental): Patients with ER+ or ER- DCIS regardless of histologic grade will be randomly assigned to receive one month standard dose chloroquine (500 mg/week).
  Interventions: Drug: Chloroquine Standard Dose (500mg/week); Procedure: Breast Biopsy
- Chloroquine Low Dose (250mg/week) (Experimental): Patients with ER+ or ER- DCIS regardless of histologic grade will be randomly assigned to receive one month low dose chloroquine (250mg/week).
  Interventions: Drug: Chloroquine Low Dose (250mg/week); Procedure: Breast Biopsy

INTERVENTIONS:
Drug: Chloroquine Standard Dose (500mg/week) — Patients will receive chloroquine (500 mg/once a week) for 1 month prior to surgical removal of the DCIS lesion.
  Other Names: Aralen
  Arms: Chloroquine Standard Dose (500mg/week)
Drug: Chloroquine Low Dose (250mg/week) — Patients will receive chloroquine (250 mg/once a week) for 1 month prior to surgical removal of the DCIS lesion.
  Other Names: Aralen
  Arms: Chloroquine Low Dose (250mg/week)
Procedure: Breast Biopsy — Patients diagnosed with DCIS will undergo a breast biopsy prior to the start of study treatment. This biopsy is entirely voluntary and is not required to remain in the study. The biopsy will allow researchers to study the tissue for biomarkers and to determine how the DCIS tissue changes during treatment. Additional samples of the DCIS tissue will be collected at the time of surgery.
  Other Names: Biopsy; DCIS; Ductal Carcinoma in Situ

SUMMARY:
The purpose of this study is to test the hypothesis that chloroquine will reduce the ability of ductal carcinoma in situ (DCIS) to survive and spread. Participants will receive either chloroquine standard dose (500mg/week) or chloroquine low dose (250mg/week) for 1 month prior to surgical removal of the tumor.

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that inhibiting the autophagy pathway in DCIS will reduce the capacity of DCIS to survive and invade. The study will examine the safety and effectiveness of neoadjuvant chloroquine administration for a one month period to patients with low, intermediate grade, or high grade DCIS. We will evaluate whether this treatment will reduce the capacity of DCIS neoplastic cells, existing within the duct, to survive, induce lesion regression, and kill the invasive DCIS progenitor cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a tissue diagnosis of low, intermediate or high grade ductal carcinoma in situ or ductal carcinoma in situ with microinvasion.
* Patients with ductal carcinoma in situ undergoing either lumpectomy/radiation or mastectomy.
* Patients must be female at least 18 years of age.
* Patients must have a signed tissue acquisition consent and have at minimum, adequate samples of primary fresh tissue or blood available for use in this study.
* No history of a previous invasive cancer in the last five years with the exception of minimally invasive non-melanoma skin cancer.
* Normal liver function based on Liver Function Tests (Total Bilirubin and Asparate transaminase (AST) <1.5 X Upper Limit of Normal).
* Normal White Blood Count (WBC) (3.5-10.8 x 103µL), Platelet count (PLT) (140-400 x 103µL), and Hematocrit (HCT)(37-52%)
* Potassium within the normal range of 3.5-5.3 mEq/L
* Adequate renal sufficiency (serum creatinine <1.5 mg/dL).
* Eastern Cooperative Oncology Group performance status 0-2.
* Are able to swallow and retain oral medication.
* No underlying ocular/retinal pathology.
* No medically documented preexisting auditory damage.
* Subjects should be willing to abstain from use of hormonal therapies (e.g. hormone replacement therapy, oral contraceptive pills, hormone-containing Intra Uterine Device (IUD)s, and E-string) and chronic non-steroidal anti-inflammatory (NSAID) s for the duration of the study (chronic use of NSAID's is defined as a frequency >3 times/week for more than two weeks per year and includes low dose aspirin).
* Subjects with child-bearing potential must agree to use adequate contraception (total abstinence (no sexual intercourse), use of condom with spermicide or sterilization surgery, including tubal ligation (tubes tied) or hysterectomy (removal of the uterus or womb)) prior to study entry and for the duration of study treatment phase. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately.

If a subject is of child-bearing potential (women are considered not of child-bearing potential if they are at least one year postmenopausal and/or surgically sterile), she must have a documented negative serum or urine pregnancy test before starting treatment.

Exclusion Criteria:

* Patients with a prior history of chemotherapy, hormonal ablation therapy and/or radiation therapy.
* History of other invasive cancer in the previous 5 years other than minimally invasive non-melanoma skin cancer.
* Patient desires not to participate in the study.
* Inability to consent.
* Current or recent pregnancy (within 12 months),
* Current use of hormone-containing forms of birth control such as implants (i.e. Norplants, or injectables ( i.e. depo-provera)
* Currently lactating.
* Patients with history of renal or hepatic insufficiency.
* Current diagnosis for depression, including treatment with an Selective Serotonin Reuptake Inhibitor (SSRI).
* History of prior treatment with chloroquine for malaria within past 24 months.
* History of allergic reactions to quinolones or chloroquine.
* Active diagnosis of psoriasis or currently receiving treatment for psoriasis.
* History of porphyria.
* History of known Glucose-6-Phosphate Dehydrogenase (G-6-PD) deficiency.
* Alcoholism or hepatic disease.
* History of epilepsy or seizures in the past 20 years.
* History of deep vein thrombosis or pulmonary embolism.
* History of human immunodeficiency virus (HIV) disease and/or treatment with anti-HIV agents.
* Receiving concurrent treatment with prohibited medications (refer to Table 1 for details on prohibited medications); Examples include: ampicillin, antacids, cimetidine, cyclosporine, kaolin, magnesium trisilicate, coumarin-type anticoagulants, macrolide antibiotics (e.g., clarithromycin, isoniazid, and erythromycin), anti-HIV agents (e.g., ritonavir and delavirdine), antidepressants (e.g. fluoxetine and fluvoxamine), calcium channel blockers (e.g. verapamil and diltiazem), steroids and their modulators (e.g., gestodene, raloxifene, and mifepristone), and several herbal and dietary components (e.g. bergamottin and glabridin).
* Used an investigational drug within 30 days or 5 half-lives, whichever is longer, preceding the first dose of study medication.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten H Edmiston, MD, FACS, Principal Investigator — Inova Fairfax Hospital Cancer Center; Priscilla McAuliffe, MD, PhD, Principal Investigator — Magee-Women's Hospital of UPMC
Locations (4):
- United States (4):
  - Medical Oncology and Hematology Associates of Northern Virginia, Fairfax, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Virginia Surgery Associates, Fairfax, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia

REFERENCES:
- [Derived] Martinez-Outschoorn UE, Pavlides S, Whitaker-Menezes D, Daumer KM, Milliman JN, Chiavarina B, Migneco G, Witkiewicz AK, Martinez-Cantarin MP, Flomenberg N, Howell A, Pestell RG, Lisanti MP, Sotgia F. Tumor cells induce the cancer associated fibroblast phenotype via caveolin-1 degradation: implications for breast cancer and DCIS therapy with autophagy inhibitors. Cell Cycle. 2010 Jun 15;9(12):2423-33. doi: 10.4161/cc.9.12.12048. Epub 2010 Jun 15. PMID 20562526

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Chloroquine Standard Dose (500mg/Week) | Chloroquine Low Dose (250mg/Week)
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chloroquine Standard Dose (500mg/Week) | Chloroquine Low Dose (250mg/Week) | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (6.6) | 56 (11.7) | 58 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 4 | 10
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 5 | 10
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Average Change in the Longest Diameter of the Breast MRI Target Lesion
Description: One of the primary outcomes of this study was to measure the impact of weekly chloroquine on the amount of DCIS seen on MRI.The tumor response was evaluated by RECIST criteria. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR The longest diameter of the target lesion or primary area of non-mass enhancement was measured by digital calipers. For one patient, the longest diameter was difficult to measure due to the presence of a significant post biopsy resolving hematoma at the biopsy site. Further correlation was made based on the extent of the pre-treatment microcalcifications and post treatment areas of non-mass enhancement.
Time Frame: Immediately preceding study drug treatment and again after treatment prior to surgery. The total time interval was up to 8 weeks
Population: The analysis population was the number of patients who underwent breast MRI both before and after treatment with chloroquine. (11/12 patients). The population was then further reduced to 10/12 due to the patient with a significant post biopsy hematoma. The extent of the pre-treatment DCIS could not be directly compared due to the presence of a significant hematoma.
Measure: Mean (Standard Deviation); unit: percentage length change
Arm/Group | Chloroquine Standard Dose (500mg/Week) | Chloroquine Low Dose (250mg/Week)
Number analyzed (Participants) | 5 | 5
percentage length change | 6 (19.8) | 43 (39)

2. Secondary Outcome: Total Number of Treatment-Related Adverse Events
Description: One of the outcomes was to ensure the safety of weekly chloroquine. Patients were followed clinically during the treatment with chloroquine and during their surgery and postoperative period ( including radiation therapy). Patients were verbally assessed for additional symptoms or concerns. Patients were also examined by the provider during treatment and follow up visits to the surgeon.
Time Frame: The patients were monitored from the time of diagnosis through 6 months of surgical follow up.
Population: Patients who were treated
Measure: Number; unit: Adverse Events (mortality, SAE, AE)
Arm/Group | Chloroquine Standard Dose (500mg/Week) | Chloroquine Low Dose (250mg/Week)
Number analyzed (Participants) | 7 | 5
Adverse Events (mortality, SAE, AE) | 0 | 0

3. Secondary Outcome: Effect of Chloroquine on Proliferating Cell Nuclear Antigen (PCNA) Proliferation Index
Description: We evaluated the effect of therapy on cellular proliferation as measured by the change in proliferating cell nuclear antigen (PCNA) proliferation index. PCNA , which is elevated during the G1/S phase of the cell cycle, may be used as a marker of cellular proliferation. The PCNA proliferation index was measured as the number of PCNA positive stained cells in the DCIS lesion/ total number of cells in the lesion. The change in the PCNA index is equal to the mean PCNA proliferation index pre-treatment minus the mean PCNA proliferation index post-treatment.
Time Frame: At the time of breast biopsy and again at time of surgery.
Population: The groups were divided by chloroquine dose. Data was only available for 6 out of 12 patients.
Measure: Mean (Standard Error); unit: Change in PCNA proliferation index
Arm/Group | Chloroquine Standard Dose (500mg/Week) | Chloroquine Low Dose (250mg/Week)
Number analyzed (Participants) | 4 | 2
Change in PCNA proliferation index | 50.4 (7.85) | 56.71 (8.11)

4. Secondary Outcome: Impact of Chloroquine Treatment on the Cell Signaling Kinase Levels in DCIS Lesions.
Description: The study evaluated the effect of chloroquine treatment on the proteomic signaling profiles of the DCIS lesions. Post treatment surgical specimens were evaluated by immunohistochemical staining to measure cell signaling kinase levels for CD68 and HMGB1. CD68 (Cluster Determinant 68) is a marker of macrophages/monocytes in the breast ducts. and HMGB1 (High Mobility Group Box 1) is involved in oxidative stress-mediated autophagy. HMGB1 is a non-histone DNA binding protein. The number of positive cells were quantified and recorded.
  .
Time Frame: At the time of surgery
Population: The analysis was performed stratifying chloroquine dose.
Measure: Mean (Standard Deviation); unit: Positive cells
Arm/Group | Chloroquine Standard Dose (500mg/Week) | Chloroquine Low Dose (250mg/Week)
Number analyzed (Participants) | 7 | 5
Positive cells
  HMGB1 | 33.9 (27.62) | 47.89 (37.99)
  CD68 | 318.3 (172.3) | 163.2 (98.2)

ADVERSE EVENTS:
Time Frame: The adverse event data was collected from the time that the chloroquin was initiated until 6 months after surgery.
Description: The definitions of adverse events was consistent with the clinicaltrials.gov definitions.
Arm/Group | Chloroquine Standard Dose (500mg/Week) | Chloroquine Low Dose (250mg/Week)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes